CLINICAL TRIAL: NCT03453021
Title: Effet du Mepolizumab Sur la décroissance de la corticothérapie systémique Chez Des Patients Avec un Asthme éosinophilique sévère Etude Observationnelle, Suivi de Cohorte Via Une ATU Nominative
Brief Title: Effect of Mepolizumab on Decrease of Systemic Corticosteroids in Patients With Severe Eosinophilic Asthma
Acronym: Mepolizumab
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC16.137
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Asthma; Eosinophilic
Keywords: asthma; mepolizumab; corticosteroids
MeSH Terms: conditions — Pulmonary Eosinophilia; Asthma | interventions — mepolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 13 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- mepolizumab: Patients will receive a subcutaneous injection of mepolizumab 100 mg every 4 weeks for one year, for a total of 12 injections
  Interventions: Drug: Mepolizumab

INTERVENTIONS:
Drug: Mepolizumab

SUMMARY:
The primary objective of the study is to measure the effect of mepolizumab on declines in oral corticosteroid therapy (prednisolone or prednisone) in patients with severe eosinophilic asthma.

Asthma is a chronic inflammatory disease of the airways that affects 5 to 10% of adults and children. Despite current treatments that are often effective, 10% of patients are not controlled by inhaled therapies. These severe asthma require regular use of systemic corticosteroids in 30 to 40% of cases. In this context, the use of glucocorticoids is associated with many more or less serious adverse effects, but still affecting the patient's quality of life. Several treatments have already been proven to save systemic steroids (theophylline, anti-leukotrienes, golimumab ...). On the other hand, none is currently recommended because of a risk / benefit ratio that is too high.

Mepolizumab is a human monoclonal antibody that binds to and inactivates interleukin 5. It has recently been shown to be effective in reducing the daily dose of oral corticosteroids and in reducing exacerbations in these patients with severe eosinophilic asthma. It also reduces the number of eosinophils in the blood and sputum and improves the quality of life.

Patients will receive a subcutaneous injection of 100mg mepolizumab every 4 weeks for one year, for a total of 12 injections.

In France, this treatment was subject to a Temporary Authorization for Nominative Use in severe eosinophilic asthma and is reserved for hospital use.

The injections will be done in HDJ Pneumology CHU Grenoble Alpes and patients will be followed monthly during injections and one month after the end of injections.

ELIGIBILITY:
Inclusion Criteria:

* Severe eosinophilic asthma
* Patient on inhaled therapy with inhaled corticosteroid and long-acting bronchodilator for at least 6 months
* Patient under oral corticosteroid therapy (prednisolone or prednisone) for at least 6 months and unmodified in the last 4 weeks before the first injection
* Patient able to provide informed and written consent
* Obtaining the temporary authorization for nominative use for mepolizumab

Exclusion Criteria:

* Chronic pulmonary pathology other than asthma
* Active neoplasia
* Active liver disease
* Serious and uncontrolled cardiovascular pathology (LVEF less than 30%, NYHA IV, ...)
* Other eosinophilic pathology (Churg & Strauss syndrome, parasitic infection, ...)
* Hypersensitivity to mepolizumab or excipient
* Immunity disorders
* Patient not affiliated to a social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included are those who have obtained the temporary authorization for nominative use for mepolizumab
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2016-01-25 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Effect of mepolizumab on declines in oral corticosteroid therapy (prednisolone or prednisone) in patients with severe eosinophilic asthma. | 13 months
  Rate of decrease in systemic corticosteroids between the day of the first injection and one month after the last injection.

SECONDARY OUTCOMES:
Asthma control | Every month during 13 months
  Asthma Control Questionnaire (ACT)
Improving quality of life | Every month during 13 months
  Asthma Quality of Life Questionnaire (AQLQ)
Improvement of respiratory functional explorations, Forced Expiratory Volume | Every month during 13 months
  Forced Expiratory Volume
Decrease in the number of exacerbations | Assessed every month during 13 months
  An exacerbation is defined as an episode of progressive degradation, over a few days, of one or more clinical signs, as well as functional parameters of bronchial obstruction.
Improvement of respiratory functional explorations | Every month during 13 months
  Vital Capacity
Improvement of respiratory functional explorations | Every month during 13 months
  Forced Vital Capacity
Improvement of respiratory functional explorations | Every month during 13 months
  FEV/FVC

CONTACTS AND LOCATIONS:
Overall Officials: Margaux Isnard, Resident, Study Chair — University Hospital, Grenoble; Laure Geneletti, Resident, Study Chair — University Hospital, Grenoble; Audrey Lehmann, Ph, Study Chair — University Hospital, Grenoble; Pierrick Bedouch, PhD, Study Chair — University Hospital, Grenoble; Sébastien Chanoine, Study Chair — University Hospital, Grenoble
Locations (1):
- University Hospital Grenoble, La Tronche, France

REFERENCES:
- [Background] Bel EH, Wenzel SE, Thompson PJ, Prazma CM, Keene ON, Yancey SW, Ortega HG, Pavord ID; SIRIUS Investigators. Oral glucocorticoid-sparing effect of mepolizumab in eosinophilic asthma. N Engl J Med. 2014 Sep 25;371(13):1189-97. doi: 10.1056/NEJMoa1403291. Epub 2014 Sep 8. PMID 25199060
- [Background] Ortega HG, Liu MC, Pavord ID, Brusselle GG, FitzGerald JM, Chetta A, Humbert M, Katz LE, Keene ON, Yancey SW, Chanez P; MENSA Investigators. Mepolizumab treatment in patients with severe eosinophilic asthma. N Engl J Med. 2014 Sep 25;371(13):1198-207. doi: 10.1056/NEJMoa1403290. Epub 2014 Sep 8. PMID 25199059